CLINICAL TRIAL: NCT04306601
Title: A Prospective, Open-Label, Single-Arm, Single-Center, Explorative Clinical Trial to Assess the Effect and Safety of Low-Intensity Focused Ultrasound on Individuals With Disorder of Consciousness After Traumatic Brain Injury
Brief Title: Low-Intensity Focused Ultrasound on Individuals With Disorder of Consciousness of Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Byung-Mo Oh, Principal Investigator Byung-Mo Oh, MD, PhD, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBI_DoC_tFUS
Record Dates: First submitted 2020-03-08; First posted 2020-03-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Traumatic Brain Injury With Prolonged Loss of Consciousness

STUDY DESIGN:
Intervention Model Description: Patients with unwakefulness syndrome or minimally conscious state after traumatic brain injury
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Intensity focused ultrasound brain stimulation (Experimental): Low-intensity focused ultrasound brain stimulation using focused ultrasound system (NS-US100; NEUROSONA Co. Ltd., Seoul, Korea)
  Interventions: Device: Low-Intensity Focused Ultrasound

INTERVENTIONS:
Device: Low-Intensity Focused Ultrasound — Low-intensity focused ultrasound brain stimulation using focused ultrasound system (NS-US100; NEUROSONA Co. Ltd., Seoul, Korea)

SUMMARY:
Low-intensity focused ultrasound can be effective in severe TBI patients with disorder of consciousness. This study is a prospective single arm, open-label and explorative clinical trial to evaluate the therapeutic effect of recovery from DoC and safety of low-intensity focused ultrasound stimulation at thalamic area in patients with post-traumatic DoC.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is an important global health concern. It is estimated that about 70 million individuals will suffer a traumatic brain injury (TBI) each year. Serious TBIs for hospitalization or death is at least 10 million annually.

Recently, advances in neurocritical care have led to an increase in the number of severe TBI patients recovering cognitive and physical function, eventually returning to independent life. However, some of severe TBI patients fail to fully recover consciousness. This condition is called disorder of consciousness (DoC). They recover from coma and maintain sleep-wake cycle, but have impaired awareness of themselves and their environment. These states are called unresponsive wakefulness syndrome or minimally conscious state. These conditions make patients loss all autonomy and heavy emotional and financial burden on their families. In addition to these devastating effects, these conditions are known to increase burn out rates in caregivers.

In the past, patients with post-traumatic DoC were considered to be "nothing to do". However, treatments such as sensory stimulation, physiotherapy, and medication have been used and studied recently. Sensory stimulation is based on the idea that enriched stimulations benefit neural plasticity and recovery. Most studies of sensory stimulation have been case-reports, with few randomized controlled study. Physiotherapy mainly includes range of motion, posture changes, and so on. Almost all hospitals offer physiotherapy, but there is still insufficient evidence to conclude that it is effective for patients with post-traumatic DoC. Studies on pharmacologic treatments in patients with DoC are mainly related to dopaminergics, because dopaminergics can stimulate the reticular activating system to improve wakefulness and attention. Among them, amantadine is proved to be an effective treatment through a large randomized controlled clinical trial in patients with post-traumatic DoC. However, although amantadine is effective in accelerating the pace of recovery, there is a limitation that the effect on long-term outcomes remains unknown.

As a scientific understanding of the consciousness grows, many studies have been conducted to restore the consciousness by neuromodulation techniques, such as median nerve stimulation, dorsal column stimulation, transcranial direct current stimulation (tDCS), repetitive transcranial magnetic stimulation (rTMS) and deep brain stimulation (DBS). Median nerve stimulation was attempted to direct sensory stimulation to the brain. However, it has been shown to be ineffective in small randomized controlled study. Attempts to stimulate the dorsal column of spinal cord directly have been made. However, because it is invasive procedure, no randomized controlled studies have been performed.

Over the past 10 years, as a restorative treatment of consciousness after TBI, the neurostimulation such as tDCS, rTMS and DBS has received increased attention. In a double-blind sham-controlled crossover design study, Thibaut et al. have investigated the efficacy of tDCS in 55 DOC patients. Significant behavioral changes were observed after tDCS in MCS patients, but after 1 year, the effect was not maintained. DBS has been generally used in Parkinson's disease, but it has been also performed in patients with DoC because it can directly stimulate thalamus. Improved the consciousness after DBS have been reported , but the evidence isn't still sufficient and the risk is too high to be administered to patients with post-traumatic DoC.

Low-intensity focused ultrasound (LIFU) has been newly proposed as a technique to overcome the limitations of existing neurostimulation techniques. LIFU has a spatial resolution of only 2-5 mm and a depth of penetration of more than 10-15 cm. Thus, it can pass through the skull to stimulate the deep brain tissue and can also stimulate finely.

In recent years, we have focused on studies of stimulating nerve tissue using a focused ultrasound stimulation system. It was reported that activation and inhibition control of motor and visual nervous system in rabbits can be achieved using a focused ultrasound stimulation system. We also reported that the thalamus of anesthetized rats was stimulated with a focused ultrasound stimulation system, resulting in a shorter recovery time from anesthesia. The image-guided navigation system using MRI made it possible to focus the ultrasound stimulation at the target point of the brain with high accuracy. In 2018, a wearable FUS headgear for a rat model was developed and the effect of long- term changes of brain function by focused ultrasound stimulation was reported, thereby identifying the possibility of neuroplasticity using LIFU.

In 2016, Monti et al. reported a clinical case of recovery of consciousness in a traffic accident patient who had been in a coma for about 20 days. The central thalamic area of the patient was stimulated with LIFU for 5-10 minutes each day, restoring consciousness from the 3rd day and starting walking on the 5th day. This result is supported by the relationship between central thalamus and consciousness. In addition, it is similar to the case that central thalamus stimulation using DBS in the patient who had MCS for 6 years after TBI modulated behavioral responses of the patient.

Based on above results, this study's aim is to evaluate the therapeutic effect of recovery from DoC and safety of LIFU stimulation at thalamic area in patients with post-traumatic DoC.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 19 years or higher
2. The patient was diagnosed with traumatic brain injury
3. A patient 6 months after brain damage
4. A patient was diagnosed with unwakefulness syndrome or minimally conscious state

Exclusion Criteria:

1. The patient needs changes of drugs that can affect changes in consciousness during the study's participation.

   * The drugs listed below are not allowed to be used in combination, unless they are being taken stably from 4 weeks prior to screening.
   * Benzodiazepines
   * Anti-epileptic drugs
   * Selective serotonin reuptake inhibitor
   * Opioids
2. Cardiopulmonary resuscitation was performed on the patient for more than 10 minutes
3. The patients has uncontrolled seizure.
4. The patient has severe thalamic atrophy of both sides, and it is impossible to determine the target area to be stimulated by sonication
5. The patient has severe medical conditions which can affect the consciousness
6. In brain computed tomography, calcification or foreign object (metallic materials, shunt catheter, etc.) that affects sonication are found in brain or skull.
7. In brain MRI, an abnormal brain blood flow or blood vessel is found
8. The patient is pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation | 6 weeks
  Coma Recovery scale - Revised
  The CRS consists of 25 hierarchically arranged items that comprise 6 subscales addressing auditory, visual, motor, oromotor, communication, and arousal processes. Scoring is based on the presence or absence of specific behavioral responses to sensory stimuli administered in a standardized manner. The lowest item on each subscale represents reflexive activity, whereas the highest items represent cognitively mediated behaviors.
  The total minimum and maximum values are 0 and 23.
Quantitative electroencephalography | 2 weeks
  Weighted phase lag index
Resting state functional MRI | 2 weeks
  ALFF (amplitude of low-frequency fluctuation)

SECONDARY OUTCOMES:
Adverse reaction | 2 weeks
  Seizure event, Electroencephalography
Rancho Los Amigos Levels of Cognitive Functioning Scale (LOCF) | 6 weeks
  Clinical evaluation of cognitive and behavioral patterns of traumatic brain injury patients
  After being assessed based on the LOCF, individuals with brain injury receive a score from one to eight. A score of one represents non-responsive cognitive functioning, whereas a score of eight represents purposeful and appropriate functioning.
Glasgow Coma Scale | 6 weeks
  Clinical evaluation of impairment of consciousness
  A person is assessed against the criteria of this scale, and the resulting points give a person's score between 3 (indicating deep unconsciousness) and either 14 (original scale) or 15 (more widely used, modified or revised scale).
Glasgow Outcome Scale Extended | 6 weeks
  The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of eight categories.
  (Death, Vegetative state, Lower severe disability, Upper severe disability, Lower moderate disability, Upper moderate disability, Lower good recovery, Upper good recovery)
  The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Mo Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data can be shared on reasonable request